CLINICAL TRIAL: NCT07219498
Title: Effects of a 5-Week Probiotic Supplementation Intervention on Markers of Delayed Onset Muscle Soreness
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Probiotic Supplementation
Record Dates: First submitted 2025-10-17; First posted 2025-10-22 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Exercise Induced Muscle Damage; Delayed Onset Muscle Soreness (DOMS)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic Group (Active Comparator)
  Interventions: Dietary Supplement: Lactobacillus casei
- Placebo Group (Placebo Comparator)
  Interventions: Other: Placebo Capsule(s)

INTERVENTIONS:
Dietary Supplement: Lactobacillus casei — Probiohealth is the manufacturer of this strain and they use a stringent quality control program that utilizes a multi point product variability check system.
  Arms: Probiotic Group
Other: Placebo Capsule(s) — The brand name of placebo capsules that will be used in this study is Magic Bullet Placebo Capsules. This placebo is manufactured by Progressive Placebo as stated on the product label.
  Arms: Placebo Group

SUMMARY:
The purpose of this study is to evaluate how probiotic supplementation (PS) influences post-exercise recovery in healthy, physically active young adults. Researchers aim to determine if the Lactobacillus casei probiotic strain reduces symptoms of delayed onset muscle soreness (DOMS) based on perceived muscle soreness, pressure pain threshold, and power output following exercise induced muscle damage (EIMD).

ELIGIBILITY:
Inclusion Criteria:

* complete a minimum of 150 minutes a week of at least moderate intensity exercise in either an endurance-based or resistance-based training style based on a self-reported physical activity over the past month
* good general health with no injuries or health conditions that would affect physical activity
* willing to abstain from consistent NSAID use and other probiotic supplements over the course of this study

Exclusion Criteria:

* known musculoskeletal injuries or physical limitations that could interfere with performing the designated physical activity required
* underlying conditions that could place them at an increased risk during exercise such as cardiovascular, respiratory, or metabolic diseases
* currently take a probiotic supplement, are prescribed and taking an antibiotic during the intervention, or report using NSAIDs or steroids within the recovery time window
* report using an NSAID more than twice a week on a regular basis

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-02-05 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in perceived muscle soreness | From baseline to post 5-week intervention
  Visual Analog Scale for perceived muscle soreness Each number on the scale will be designated with a descriptive word that corresponds to the soreness level they are experiencing. The scale will be laid out in order of increasing muscle soreness with "1" representing no pain.
Change in pressure pain threshold (PPT) | From baseline to post 5-week intervention
  Calf pressure pain threshold (PPT) will be assessed by placing marks on the medial condyle of the femur and the posterior of the medial malleolus. The researcher will place the algometer on the muscle belly exactly halfway between the two marks. Volunteers will be instructed to specify when the first onset of pain occurs as the researcher gradually applies pressure. Quadricep measurements will involve the participant lying in the supine position where marks will be made on the anterior inferior iliac spine and the top of the patella so the researchers can once again find a point exactly halfway between these two locations to apply the algometer. Participants will be instructed to verbally indicate to the researcher when the onset of pain occurs as pressure is applied.
Change in countermovement jump assessment (CMJ) performance recovery | From baseline to post 5-week intervention
  The researchers will demonstrate and instruct volunteers to "Stand upright with their hands above their head. When you are ready, bend your knees and stick your hips back while keeping your hands to your hips. Jump as high as possible and land softly." Participants will perform three CMJs separated by 60 seconds. Jump height will be recorded in cm and the highest value will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Stenson, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No